CLINICAL TRIAL: NCT02407808
Title: Cannabinoids, Learning, and Memory
Acronym: THC-Memory
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Associate Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1501015211; No NIH funding (Other: 10.11.23)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cannabis; Psychotic Disorders
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- THC (Active Comparator): Active THC (0.0015mg/kg-0.03mg/kg) administered over 20 minutes.
  Interventions: Drug: THC; Drug: Placebo
- Placebo (Placebo Comparator): Control: small amount of alcohol intravenously (quarter teaspoon), with no THC over 20 minutes.
  Interventions: Drug: THC; Drug: Placebo

INTERVENTIONS:
Drug: THC — Active THC (0.0015-0.03 mg/kg) administered over 20 minutes.
Drug: Placebo — Control: small amount of alcohol intravenously (quarter teaspoon), with no THC over 20 minutes.

SUMMARY:
The overarching goal of this study is to characterize the effects of cannabinoids on working and episodic memory.

DETAILED DESCRIPTION:
This study will be achieved by studying the acute effects of delta-9-tetrahydrocannabinol (THC), the main psychoactive component of cannabis and a cannabinoid-1 receptor (CB1R) agonist, on a wide range of memory tasks in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and 55 years (extremes included) on day of first dosing
* Exposed to cannabis at least once in their lifetime

Exclusion Criteria:

* Cannabis naive
* Positive pregnancy screen during screening
* Hearing deficits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-08-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Test (RAVLT) | +35 minutes after infusion
  a measure of verbal episodic memory
N-Back Task | +65 minutes after infusion
  a measure of working memory

SECONDARY OUTCOMES:
Clinician Administered Dissociative Symptoms Scale (Total Score) | Baseline, +10, +85, and +240 minutes after the first infusion
Visual Analog Scale (Total Score) | Baseline, +10, +85, +240 minutes after the first infusion
  a measure of THC intoxication

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, M.D., Principal Investigator — Assistant Professor
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States